CLINICAL TRIAL: NCT01999010
Title: Mental Health Telemetry for Self-Management in Major Depression
Acronym: MHTV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 186-2013
Record Dates: First submitted 2013-08-01; First posted 2013-12-03 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder
Keywords: psychiatry; mental health; major depressive disorder; self-management; data visualization; mood diaries; electronic diaries; cell phones; software; mental health telemetry; ecological momentary assessment
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment as usual ("A" Stage) (No Intervention): The treatment as usual (TAU) group will continue to receive their usual treatment from their current treatment team - i.e. MHT will not be introduced during this phase.
- MHT ("B" Stage) (Experimental): Patients will be given software for Mental Health Telemetry (MHT), which allows them to record symptom intensity, hospital / ER visits, life events, etc., and to visualize their MHT data. Patients will be encouraged to make MHT entries once daily at a pre-determined time while in this arm, and will be prompted via text message by the MHT software to do so.
  Interventions: Device: MHT
- Choice ("A' " Stage) (Experimental): Patients exiting the MHT arm will be given the choice to continue with MHT for a further two months or whether to resume TAU (i.e., no further use of MHT) for the remaining two months.
  Interventions: Device: MHT

INTERVENTIONS:
Device: MHT — MHT and visualizer contains mood information about the patient themselves, which allows for self management of the mood disorder. Self-management interventions promote early recognition of mood episodes, medication adherence and self-management skills which have shown to improve outcomes in depression. MHT encourages patients to take an active role by engaging in mood journaling, while making this information available in explorable form to the patient and his / her team of clinicians.
  Arms: Choice ("A' " Stage); MHT ("B" Stage)

SUMMARY:
Mood journaling is a cornerstone of self-management in major depressive disorder (MDD). Research over the last decade has shown that electronic mood journals are superior to paper ones. One potential advantage of mental health telemetry (MHT), which use cell phones to collect mood journal data, is that electronic journal data can easily be converted into graphical records, allowing people living with MDD to readily spot trends, correlations, or patterns in ways that would be quite challenging using paper diaries. This information should make it easier to recognize and evaluate changes in mental health status -- the first two steps in the process of self-management. The investigators will develop and deploy a visualization module for patients with which to explore their own MHT data sets on the same cell phones which they record their journals, and test the investigators hypotheses that their enhanced MHT system will (i) improve patients' ability to self-manage MDD and (ii) enhance their quality-of-life.

The study is a non-randomized, un-blinded, A-B-A' (modified single-subject withdrawal design, with user choice of treatment or withdrawal in the A' stage) study, to explore the utility of MHT as a tool for enhancing self-management and QoL for persons living with MDD. The aims of this study are to explore the impact of MHT on subjects' self-management and QoL, and to gauge participants' perceptions of MHT's utility.

ELIGIBILITY:
We will recruit (n=113) patients with a Diagnostic and Statistical Manual, 4th Ed. (DSM-IV) diagnosis of MDD, confirmed using the MDD section of the M.I.N.I. International Neuropsychiatric Interview (MINI) version 5.0. All recruits will own or use a web-enabled cell phone.

Exclusion Criteria:

* self-disclosed illiteracy;
* blindness;
* inability to be successfully trained in the use of MHT

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in self-management ratings | two months and four months
  Self-management ratings using the three sub-scale scores (maintenance, management, and confidence) of the Sunnybrook Self-Management Scale - Depression (3S-D) instrument at the end of the Treatment-as-Usual phase (two months) as compared to the end of the active treatment phase (four months)

SECONDARY OUTCOMES:
Change in Quality-of-life (QoL) ratings | two months and four months
  Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ) scores at the end of the treatment-as-usual (two months) and active treatment (four months) phases. We will control for severity of mood symptoms (using mental health telemetry (MHT) composite depression scores) as a covariate of the magnitude of change in QoL outcomes because we expect that some, but not all, of the variance in QoL outcomes will be accounted for in particular by the severity of depression.

OTHER OUTCOMES:
Retention Rates (Exploratory) | Four months
  We will report the proportion and 95% confidence interval (CI) of users who opt to continue using MHT in the A' (user choice) phase
Utilization Rates (Exploratory) | Six months
  We will report the mean number and 95% CI of times per patient (in the B and A' phases) that MHT data was (i) reported and (ii) visualized.

CONTACTS AND LOCATIONS:
Overall Officials: David M Kreindler, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada